CLINICAL TRIAL: NCT00565708
Title: Aspirin for Dukes C and High Risk Dukes B Colorectal Cancers - An International, Multi-Center, Double Blind, Randomized Placebo Controlled Phase III Trial
Brief Title: Aspirin for Dukes C and High Risk Dukes B Colorectal Cancers
Acronym: ASCOLT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Centre, Singapore (Other)
Collaborators: Australasian Gastro-Intestinal Trials Group (Network); INDOX Cancer Research Network (Other); University of Sydney (Other)
Responsible Party: Principal Investigator, Toh Han Chong, Prof, National Cancer Centre, Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CDR0000577892; SINGAPORE-ICR-02 (Other: SCRI); SINGAPORE-ASCOLT (Other: SCRI)
Record Dates: First submitted 2007-11-29; First posted 2007-11-30 (Estimated); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Colorectal Cancer
Keywords: stage II colon cancer; stage III colon cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acetylsalicylic acid (Experimental): 200mg OD for 3 years
  Interventions: Drug: Acetylsalicylic acid
- Placebo (Placebo Comparator): 200mg OD for 3 years
  Interventions: Other: placebo

INTERVENTIONS:
Other: placebo — Placebo Comparator
  Arms: Placebo
Drug: Acetylsalicylic acid — Adjuvant Therapy
  Other Names: Aspirin
  Arms: acetylsalicylic acid

SUMMARY:
We hypothesize through this randomized, placebo-controlled adjuvant study, that Aspirin in patients with dukes C or high risk dukes B colorectal cancer (ASCOLT) can improve survival in this patient population over placebo control. If indeed found to be beneficial, because aspirin is cheap and easy to administer, it will positively impact the lives of many individuals in Asia and globally.

STUDY OBJECTIVE

To assess the effectiveness of Aspirin against placebo control in patients with dukes C or high risk dukes B colorectal cancer in terms of Disease Free Survival (DFS) and Overall Survival (OS)

Primary endpoints

* DFS among all eligible subjects (high risk Dukes B colon cancer, Dukes C colon cancer and rectal cancer patient sub-groups);
* DFS among patients with colon cancer (high-risk Dukes B and Dukes C colon cancer).

Secondary endpoints

* Overall survival (OS) over 5 years
* DFS and OS in

  * Chinese, Malay, Indian and other ethnic groups
  * Resected high risk Dukes B colon cancer, Dukes C colon cancer and rectal cancer sub-groups, individually
  * Compliant versus non-compliant subjects
  * PIK3CA mutated tumors (where samples are available)

DETAILED DESCRIPTION:
Aspirin in patients with dukes C or high risk dukes B colorectal cancer can improve survival in this patient population over placebo control.

Eligible patients will be randomized to treatment arms, using the following stratification factors:

* Study Centre
* Tumour Type
* Type of adjuvant chemotherapy received(exposed/not exposed to oxaliplatin

Patients will be randomized over a 5 years' time period. After randomization, patient will have 3 monthly assessments with treatment for 3 years followed by 6 monthly assessments for additional 2 years follow-up

ELIGIBILITY:
Inclusion Criteria

* Male or female outpatient of ≥ 18 years of age or ≥ country's legal age for adult consent
* Dukes C colon cancer, high risk Dukes B colon cancer, Dukes B rectal cancer or Dukes C rectal cancer (see Appendix 1 for definition of High Risk Dukes B)
* Undergone complete resection of primary tumour
* Completed standard therapy ( at least 3 months of chemotherapy ± radiotherapy )
* Within 120 days of completion of standard therapy (surgery, chemotherapy ± radiotherapy)
* ECOG performance status 0 to 2
* Satisfactory haematological or biochemical functions (tests should be carried out within 8 weeks prior to randomisation): Results of clinical investigations carried out within 8 weeks prior to randomisation can be used in place of the required screening investigations. Patients with mild laboratory abnormalities can be included at the discretion by the site principal investigator, and after approval by ASCOLT Trial Management Group
* ANC ≥ 1.0 x 109/L
* Platelets ≥ 100 x 109/L
* Creatinine clearance ≥ 30 mL/min
* Total bilirubin ≤ 2.0 x the upper limit normal
* AST & ALT ≤ 5 x the upper limit normal
* Completed the following investigations
* Colonoscopy(or CT colonogram(within 16 months prior to randomization)
* Imaging of abdomen (CT or CT colonogram or MRI or PET or Ultrasound) within 16 months prior to randomization
* Written informed consent

Exclusion Criteria

* Pre-existing Familial adenomatous polyposis, inflammatory bowel disease or ulcerative colitis
* Active gastritis or active peptic ulcer
* History of continuous daily use of PPI more than 1 year prior to consent
* Gastrointestinal bleeding within the past one year
* Haemorrhagic diathesis (i.e. haemophilia)
* Uncontrolled hypertension (untreated systolic blood pressure > 160 mmHg, or diastolic blood pressure > 95 mmHg)
* History of recent cancers (except for colorectal cancers, non-melanoma skin cancers, basal cell carcinomas, squamous cell carcinomas) in the past 5 years
* History of stroke, coronary arterial disease, angina, or vascular disease
* Patients who are on current long term treatment (≥ 4 consecutive weeks) with Aspirin, NSAID or Cox-2 inhibitors
* History of erosive GERD or active erosive GERD on gastroscopy.
* Patient on active current treatment of antiplatelet agents (i.e. off-study Aspirin, clopidogrel, ticlopidine)
* Patient receiving active treatment of anticoagulants (i.e. warfarin, low molecular weight heparins)
* Pregnant, lactating, or not using adequate contraception
* Patient having known allergy to NSAID or Aspirin
* Unexplained rise of CEA (i.e. smoker with elevated CEA will not be excluded)
* Patient on other investigational drug
* Patients with HNPCC (Lynch Syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1587 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 5 years
  Recurrence data documented

SECONDARY OUTCOMES:
Overall survival | 5 years
  Death data documented

CONTACTS AND LOCATIONS:
Overall Officials: John Chia, MBBS, MRCP, Study Chair — National Cancer Centre, Singapore; Raghib Ali, MBBS,MRCP, Study Chair — NYU; Han Chong Toh, MD,MBBS,MRCP, Study Chair — National Cancer Centre, Singapore; Eva Segelov, MBBS,PhD, Study Chair — Monash University, University of Bern
Locations (67):
- Australia (29):
  - Bankstown-Lidcombe Hospital Bankstown Cancer Centre, Bankstown, New South Wales
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Clinical Research Centre, Camperdown, New South Wales
  - Coffs Harbour Health Campus North Coast Cancer Institute, Coffs Harbour, New South Wales
  - Central Coast Cancer Centre Gosford Hospital, Gosford, New South Wales
  - Newcastle private Hospital, New Lambton Heights, New South Wales
  - Orange Health Service, Orange, New South Wales
  - Port Macquarie Base Hospital North Coast Cancer Institute, Port Macquarie, New South Wales
  - Northern Cancer Institute, St Leonards, St Leonards, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - Northwest Cancer Centre Tamworth Hospital, Tamworth, New South Wales
  - The Tweed Hospital, Tweed Heads, New South Wales
  - Calvary Mater Newcastle Hospital, Waratah, New South Wales
  - Royal Darwin Hospital, Tiwi, Northern Territory
  - Townsville Hospital, Douglas, Queensland
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Border Medical Oncology Research Unit, Albury, Victoria
  - Ballarat Regional Integrated Cancer Centre, Ballarat, Victoria
  - Barwon Health Andrew Love Cancer Centre, Geelong, Victoria
  - Austin Health Cancer Clinical Trials, Heidelberg, Victoria
  - Launceston General Hospital, Launceston, Victoria
  - Monash Health Medical Oncology, Melbourne, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - St John of God Healthcare Southwest Oncology, Warrnambool, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - St John of God Hospital Subiaco, Subiaco, Western Australia
- China (15):
  - Beijing University Cancer Hospital, Beijing, Beijing Municipality
  - The First People's Hospital of Foshan City, Foshan, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Sixth Affiliated Hospital, Guangzhou, Guangdong
  - Sun Yat Sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan City People's Hospital, Zhongshan, Guangdong
  - Affiliated Hospital of Nantong University, Nantong, Jiangsu
  - Jinan Central Hospital, Jinan, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shuang Ho Hospital, Taibei, Taiwan
  - Koo Foundation Sun Yat Sen Cancer Centre, Taibei, Taiwan
  - Taipei Medical University Hospital, Taibei, Taiwan
  - Wan Fang Hospital, Taibei, Taiwan
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Queen Mary Hospital - Hong Kong, Hong Kong
- India (7):
  - Kidwai Memorial Institute of Oncology, Bangalore
  - G. Kuppuswamy Naidu Memorial Hospital, Coimbatore
  - Nizam's Institute of Medical Sciences, Hyderabad
  - Tata Memorial Hospital, Mumbai
  - All India Institute of Medical Sciences, New Delhi
  - Regional Cancer Center, Trivandrum
  - Christian Medical College and Hospital, Vellore
- Indonesia (3):
  - Dharmais Cancer Hospital, Jakarta
  - Cipto Mangunkusumo General Hospital, Jakarta
  - Rumah Sakit RSUP Dr. Sardjito, Yogyakarta
- Malaysia (4):
  - Sarawak General Hospital, Kuching, Sarawak
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University of Malaysia Medical Center, Kuala Lumpur
  - University Kebangsaan Malaysia Medical Center, Kuala Lumpur
- New Zealand (2):
  - Christchurch Public Hospital, Christchurch
  - Dunedin Hospital, Dunedin
- King Fahad Medical City, Riyadh, Saudi Arabia
- Singapore (3):
  - National Cancer Centre - Singapore, Singapore
  - Johns Hopkins Singapore International Medical Center, Singapore
  - Tan Tock Seng Hospital, Singapore
- South Korea (2):
  - Hallym University Sacred Heart Hospital, Anyang-si, Gyeonggi-do
  - Severance Hospital, Seoul
- National Cancer Institute, Maharagama, Sri Lanka

REFERENCES:
- [Background] Segelov E, Prenen H, Day D, Macintyre CR, Foo EMJ, Ali R, Wang Q, Wei X, Lopes GL Jr, Ding K, Chen G, Chia JWK, Toh HC; ASCOLT Investigators. Impact of the COVID-19 Epidemic on a Pan-Asian Academic Oncology Clinical Trial. JCO Glob Oncol. 2020 Apr;6:585-588. doi: 10.1200/GO.20.00072. No abstract available. PMID 32293940
- [Background] Day D, Toh HC, Ali R, Foo EMJ, Simes J, Chia JWK, Segelov E; ASCOLT Investigators. Operational Challenges of an Asia-Pacific Academic Oncology Clinical Trial. JCO Glob Oncol. 2023 Jun;9:e2300040. doi: 10.1200/GO.23.00040. PMID 37364220
- [Derived] Chia JWK, Segelov E, Deng Y, Ho GF, Wang W, Han S, Sharma A, Ding K, Chen G, Jeffery MG, Tham CK, Ahn JB, Nott L, Zielinski R, Chao TY, van Hagen T, Wei PL, Day F, Mehta S, Yau T, Peng J, Hayes TM, Li Y, Gandhi M, Foo EMJ, Rahman N, Rothwell P, Ali R, Simes J, Toh HC. Aspirin after completion of standard adjuvant therapy for colorectal cancer (ASCOLT): an international, multicentre, phase 3, randomised, double-blind, placebo-controlled trial. Lancet Gastroenterol Hepatol. 2025 Mar;10(3):198-209. doi: 10.1016/S2468-1253(24)00387-X. Epub 2025 Jan 14. PMID 39824200
- [Derived] Ali R, Toh HC, Chia WK; ASCOLT Trial Investigators. The utility of Aspirin in Dukes C and High Risk Dukes B Colorectal cancer--the ASCOLT study: study protocol for a randomized controlled trial. Trials. 2011 Dec 14;12:261. doi: 10.1186/1745-6215-12-261. PMID 22168568

DOCUMENTS (2):
  • Study Protocol (2018-05-09): https://cdn.clinicaltrials.gov/large-docs/08/NCT00565708/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/08/NCT00565708/SAP_001.pdf